CLINICAL TRIAL: NCT00032994
Title: Motivational Interviewing (MI) to Improve Treatment Engagement and Outcome in Subjects Seeking Treatment for Substance Abuse
Brief Title: Motivational Interviewing to Improve Treatment Engagement and Outcome in Subjects Seeking Treatment for Substance Abuse - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Kathleen Carroll, Ph.D., Yale University School of Medicine
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NIDA-CTN-0005-1; NCT00015730 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-04

CONDITIONS: Substance-Related Disorders
Keywords: substance use disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to assess Motivational Interviewing (MI) to improve treatment engagement and outcome in subjects seeking treatment for substance abuse.

DETAILED DESCRIPTION:
Participants seeking treatment at the participating CTPs will be randomly assigned to either "standard" or "MET/MI" treatment, with a 1- and 3-month follow-up. Primary outcome measures will include (1) treatment retention (e.g., number of sessions/weeks completed, the rate of patients completing 3 or more subsequent sessions, and (2) substance use (e.g., urinalyses, days of opioid, cocaine, marijuana, alcohol use, rates of abstinence). Secondary outcomes will include motivation, psychosocial functioning, HIV risk behaviors, treatment utilization, and patient satisfaction. Process assessments will include measures of the working alliance as well as therapist adherence/competence ratings which will evaluate how effectively MET/MI was implemented. Participating CTPs will implement one of two independent protocols, depending on which is the best suited or feasible for the intake procedures at their clinic. Thus, following an invitation to participate, explanation of the study, and provision of informed consent, patients would complete a brief assessment battery followed by either:1) Random assignment to 3 individual sessions of standard treatment (treatment as usual) at the program versus 3 individual sessions of MET; or 2) Random assignment to 1 individual standard assessment/evaluation session.

ELIGIBILITY:
Inclusion Criteria:

Individuals will be eligible for the protocol who: a)Are seeking outpatient treatment for any substance use disorder. b)Are 18 years of age or older. c)Are willing to participate in the protocol (e.g., to be randomized to treatment, be contacted for follow-up assessment, to have their sessions audiotaped). d)Are able to understand and provide written informed consent.

Exclusion Criteria:

Individuals will be excluded who: a)Are not sufficiently medically or psychiatrically stable to participate in outpatient treatment. b)Are seeking detoxification only, methadone maintenance, or residential inpatient treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422
Dates: Start 2001-04; Primary Completion 2002-10 (Actual); Study Completion 2002-10

PRIMARY OUTCOMES:
Drug use
Retention
HIV risk behaviors
Psychosocial functioning

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, Ph.D., Principal Investigator — VA Connecticut Healthcare System
Locations (5):
- United States (5):
  - Lower Eastside Service Center (LESC), New York, New York
  - Willamette Family Treatment Services, Eugene, Oregon
  - Changepoint - Cedar Hills Blvd, Portland, Oregon
  - ADAPT, Roseburg, Oregon
  - Chesterfield County CSB- Substance Abuse Services, Chesterfield, Virginia

REFERENCES:
- See also: Data Elements — http://www.ctndatashare.org/protocol-ctndatashare/new-protocols/nida-ctn-0005